CLINICAL TRIAL: NCT04537351
Title: A Pilot, Open-label, Randomised Controlled Clinical Trial to Investigate Early Efficacy of CYP-001 in Adults Admitted to Intensive Care With Respiratory Failure
Brief Title: The MEseNchymal coviD-19 Trial: MSCs in Adults With Respiratory Failure Due to COVID-19 or Another Underlying Cause
Acronym: MEND
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cynata Therapeutics Limited (Industry)
Collaborators: Cerebral Palsy Alliance (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CYP-COVID-19-01
Record Dates: First submitted 2020-08-25; First posted 2020-09-03 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Covid19; Acute Respiratory Distress Syndrome
Keywords: Mesenchymal stem cells; MSC; Induced pluripotent stem cells; iPSC; Cellular therapy
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- CYP-001 (Experimental): The investigational medicinal product used in this study is known as CYP-001. The active agent in CYP-001 is Cymerus™ MSCs. CYP-001 is supplied as 100 million Cymerus MSCs formulated in 20 mL cryoprotectant medium. On D1 and D3, each participant randomised to receive CYP-001 will receive an IV infusion of 2 million Cymerus MSCs/kg of body weight (up to a maximum of 200 million cells per infusion).
  Interventions: Biological: CYP-001
- Standard of care (No Intervention): Control participants will be randomised to received standard of care treatment.

INTERVENTIONS:
Biological: CYP-001 — The active agent in CYP-001 is Cymerus mesenchymal stem cells (MSCs), which are derived through a proprietary induced pluripotent stem cell (iPSC) and mesenchymoangioblast (MCA)-derived production process.
  Other Names: Cymerus MSCs
  Arms: CYP-001

SUMMARY:
This is a pilot, multi-centre, open-label randomised controlled study to assess the early efficacy of intravenous (IV) administration of CYP-001 in adults admitted to an intensive care unit (ICU) with respiratory failure

DETAILED DESCRIPTION:
After enrolment upon meeting eligibility criteria (D0), participants baseline data will be collected and participants will be randomised to receive either standard of care treatment only, or standard of care plus CYP-001. On D1 and D3, each participant randomised to receive CYP-001 will receive an IV infusion of 2 million Cymerus mesenchymal stem cells (MSCs)/kg of body weight (up to a maximum of 200 million cells). Participants will have further data collection throughout their ICU and hospital stay and follow up to 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older
* Respiratory failure with the following signs and symptoms:

  1. P/F ratio <300 mmHg
  2. Onset within one week of a known insult or new or worsening respiratory symptoms.
  3. Chest imaging shows bilateral opacities, which are not fully explained by effusions, lobar/lung collapse, or nodules.
* Respiratory failure which is not fully explained by cardiac failure or fluid overload.
* Onset of respiratory failure within the past 48 hours (as defined in inclusion criterion 2

Exclusion Criteria:

* <18 years of age
* Patient is known to be pregnant
* Known active malignancy that required treatment in the last year
* WHO Class III or IV pulmonary hypertension
* Venous thromboembolism currently receiving anti-coagulation or within the past 3 months
* Currently receiving extracorporeal life support
* Severe chronic liver disease (Child-Pugh score >12)
* "Do Not Attempt Resuscitation" order in place
* Treatment withdrawal imminent within 24 hours
* BMI > 45 kg/m2.
* Received any investigational research agent within 60 days or within five half-lives of the last treatment (if the half-life of the investigational agent is known to be longer than 12 days) prior to the planned administration of study treatment.
* Known positive test for human immunodeficiency virus 1 (HIV 1), HIV 2, hepatitis B virus, Hepatitis C virus or any other infection which the opinion of the Investigator is likely to impact on the ability of the patient to participate in the study.
* Known sensitivity to dimethylsulfoxide (DMSO) or any other component of the study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-05-18 (Actual)

PRIMARY OUTCOMES:
Trend in trajectory of PaO2/FiO2 ratio (P/F ratio) between groups | 7 days
  Assessment of respiratory dysfunction

SECONDARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events | 28 days
  Assessment of safety
Change in C-reactive protein (CRP) levels | 7 days
  Circulating biomarker of inflammation
Proportional differences between groups on the Clinical Improvement Scale | 28 days
  Not hospitalised, with resumption of normal activities = 1; Not hospitalised, but unable to resume normal activities = 2; Hospitalised, not requiring supplemental oxygen = 3; Hospitalised, requiring supplemental oxygen = 4; Hospitalised, requiring humidified nasal high-flow oxygen therapy, non-invasive mechanical ventilation, or both = 5; Hospitalised, requiring invasive mechanical ventilation, extracorporeal membrane oxygenation or both = 6; Death = 7
Changes in P/F ratio | 28 days
  Assessment of respiratory dysfunction
Changes in respiratory rate | 28 days
  Assessment of respiratory dysfunction
Changes in oxygenation index | 28 days
  Assessment of respiratory dysfunction
Changes in respiratory compliance (the change in lung volume per unit change in transmural pressure gradient) | 28 days
  Assessment of respiratory dysfunction
Changes in positive end-expiratory pressure | 28 days
  Assessment of respiratory dysfunction
Ventilator-free days | 28 days
  Number of days from the time of initiating unassisted breathing to D28, assuming survival for at least 48 hours after initiating unassisted breathing and continued unassisted breathing to D28
Proportional differences between groups on the SF-36 | 28 days
  Quality of life assessment
Proportional differences between groups on the mini mental state examination | 28 days
  Disability assessment

CONTACTS AND LOCATIONS:
Overall Officials: Jolanta Airey, MD, Study Director — Cynata Therapeutics Limited
Locations (5):
- Australia (5):
  - Nepean Hospital, Kingswood, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Footscray Hospital, Footscray, Victoria
  - Sunshine Hospital, Saint Albans, Victoria

IPD SHARING:
Plan to Share IPD: Yes
IPD relating to efficacy of MSCs in COVID-19 may be shared, subject to permission from Sponsor and ethics approval if required. All de-identified data collected during this study may be shared confidentially to contribute to meta-analysis of mesenchymal stem cell treatments for COVID-19. Request for IPD from this trial for other purposes will be considered by the Sponsor.
Time Frame: Data requests will be considered after the completion of the study. There is no specified end date.
Access Criteria: All reasonable requests for raw and analysed data that are not included in primary publications from this study may be available upon request and discretion from the Sponsor from the beginning to the trial. Data may be made available to active collaborators in the COVID-19 Stem Cell Treatment (CSCT) Group, subject to permission from the Sponsor and ethics approval if required. All other reasonable requests for raw and analysed data will be considered by the Sponsor. Data may be obtained upon permission from the Sponsor.